CLINICAL TRIAL: NCT05688475
Title: Continuing Treatment for Participants Who Have Participated in a Prior Protocol Investigating CC-122
Brief Title: A Rollover Study of CC-122
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA092-1000; 2022-501855-97 (EudraCT Number); U1111-1282-2472 (Registry Identifier: WHO)
Record Dates: First submitted 2023-01-10; First posted 2023-01-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: CC-122; Avadomide; BMS-986381; Non-Hodgkin Lymphoma; Diffuse large B cell lymphoma; Follicular lymphoma; Chronic lymphocytic leukemia; Multiple myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-122 and Dexamethasone (Experimental)
  Interventions: Drug: CC-122; Drug: Dexamethasone

INTERVENTIONS:
Drug: CC-122 — Specified dose on specified days
  Other Names: Avadomide; BMS-986381
Drug: Dexamethasone — Specified dose on specified days

SUMMARY:
The purpose of the study is to provide CC-122 treatment to participants who have been receiving treatment in other CC-122 clinical trials investigating CC-122 for more than 5 years (CC-122-ST-001 [NCT01421524], CC-122-ST-002 [NCT02509039], CC-122-DBCL-001 [NCT02031419], and CC-122-NHL-001 [NCT02417285]), receiving clinical benefit from the treatment and to monitor the safety and tolerability of CC-122.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant who is currently receiving CC-122 on another CC-122 clinical trial that has met its primary and secondary endpoints.
* Participant who has participated in previous CC-122 protocol (including CC-122-ST-001 [NCT01421524], CC-122-ST-002 [NCT02509039], CC-122-DBCL-001 [NCT02031419], and CC-122-NHL-001 [NCT02417285]), and is deemed by the investigator to be deriving benefit from CC-122 as defined by the previous protocol.
* Participant who is able to tolerate study therapy and has not yet experienced progressive disease or any treatment discontinuation criteria of the Parent Study.

Key Exclusion Criteria:

* Participant is not eligible for CC-122 treatment as per the Parent Study.
* Participants not receiving clinical benefit as assessed by the investigator. Any clinical AE, laboratory abnormality, or intercurrent illness which, in the opinion of the investigator, indicates that participation in the study is not in the best interest of the participant.
* Women who are breastfeeding.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious adverse events (SAEs) for participants who received at least 1 dose of CC-122 | Up to approximately 3 years
Number of deaths for participants who received at least 1 dose of CC-122 | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (3):
  - Local Institution - 100, New York, New York
  - Local Institution - 101, Nashville, Tennessee
  - Local Institution - 102, Madison, Wisconsin
- France (2):
  - Local Institution - 300, Bordeaux
  - Local Institution - 301, Marseille
- Local Institution - 500, Koto-ku, Tokyo, Japan
- Local Institution - 400, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05688475.html